CLINICAL TRIAL: NCT06757764
Title: The Effect and Safety of Therapy Adding Cilostazol in Acute Ischemic Stroke Due to Large Artery Atherosclerosis: CHANGE Trial
Brief Title: The Effect and Safety of Combined Anti-platelet Treatment in Acute Ischemic Stroke Due to Large Artery Atherosclerosis
Acronym: CHANGE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Bum Joon Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHANGE
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Infarction; Stenosis Artery
MeSH Terms: conditions — Cerebral Infarction | interventions — Aspirin; Clopidogrel; Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CA group (Experimental): Aspirin 100mg qd (21days), clopidogrel 75mg qd (180days), Cilostazol SR 100mg x 2cap (180days). In case of stenting, aspirin will be added to cilostazol and clopidogrel until 90 days after stenting.
  Interventions: Drug: Aspirin; Drug: Clopidogrel; Drug: Cilostazol
- PA group (Placebo Comparator): Aspirin 100mg (21days), clopidogrel 75mg qd (180days), Placebo x 2cap (180days). In case of stenting, aspirin will be added to placebo and clopidogrel until 90 days after stenting.
  Interventions: Drug: Aspirin; Drug: Clopidogrel; Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — Aspirin 100mg qd (21days)
  * In case of stenting, aspirin will be added to cilostazol and clopidogrel until 90 days after stenting.
  * Route: per oral. IMP can be taken with or without food.
  * Frequency: once daily (qd)
Drug: Clopidogrel — Clopidogrel 75mg qd (180days)
  * Route: per oral. IMP can be taken with or without food.
  * Frequency: once daily (qd)
Drug: Cilostazol — Cilostazol SR 100mg x 2cap (180days)
  * Route: per oral. IMP can be taken with or without food.
  * Frequency: once daily (qd)
  Arms: CA group
Drug: Placebo — Placebo x 2cap (180days)
  * Route: per oral. IMP can be taken with or without food.
  * Frequency: once daily (qd)
  Arms: PA group

SUMMARY:
Currently, aspirin plus clopidogrel is considered as a standard acute treatment of ischemic stroke, based on results of CHANCE and POINT trial. However, still a considerable portion of patients showed early stroke recurrence, especially in those with stroke due to large artery atherosclerosis. Cilostazol may have benefit in reducing early stroke recurrence of neurologic deterioriation. The post-hoc analysis of CSPS.com showed that use of cilostazol after 15 days of stroke was effective for preventing subsequent stroke. The effect of adding cilostazol was more effective in those with large artery atherosclerosis and those receiving clopidogrel than aspirin.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 20 years or older
2. Acute ischemic stroke due to large artery atherosclerosis (both including Intra and extracranial atherosclerosis) which may be defined by a ischemic lesion confirmed at diffusion-weighted image and a corresponding significant stenosis (more than 50% of diameter reduction) proximal to the ischemic lesion confirmed by MR or CT angiography.
3. Able to start IMP within 72h from stroke onset
4. Acquisition of written informed consent prior to study entry

Exclusion Criteria:

1. Large infarction unable to start antiplatelet treatment
2. Combined with acute intracranial haemorrhage
3. With initial haemorrhagic transformation
4. Previous mRS higher than 2
5. Indicated for anticoagulation
6. Contraindication for aspirin, clopidogrel or cilostazol
7. Requirement of long term NSAID
8. Pre-planned for surgery
9. Unable to withdraw consent
10. Unavailable to participate based on judgement of the investigator
11. Participants of reproductive potential (PORP)/ Participants of childbearing potential (POCBP) who do not agree to practice methods of birth control or remain fully abstinent from sexual activity with the potential for conception.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2340 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of occurrence of composite endpoint | during admission (within 14 days) and within 180 days after stroke
  *Composite endpoint: Neurologic deterioration† during admission (within 14 days) or recurrence of ischemic stroke‡ within 180 days after stroke
  †Neurologic deterioration: Increment of 2 or more in total NIHSS(National Institutes of Health Stroke Scale) score or one or more in the motor NIHSS score.
  ‡Recurrence of ischemic stroke: A newly developed neurological deficit corresponding to a new ischemic lesion confirmed by neuro-imaging.

SECONDARY OUTCOMES:
Proportion of participants with good functional outcome (mRS(modified Rankin Scale) 0-2) | at 180 days
mRS score collected at 180 days | at 180 days
Proportion of participants with Neurologic Deterioration(ND) during admission | during admission(within 14days)
Proportion of participants with good functional outcome (mRS 0-2) | at 90 days
Proportion of participants with ischemic stroke recurrence | at 90 days
Proportion of participants with ischemic stroke recurrence | at 180 days
Proportion of participants with MI(Myocardial Infarction), ischemic stroke recurrence, haemorrhagic stroke and vascular death | within 180 days
Proportion of participants with haemorrhagic stroke | within 180 days
Proportion of participants with myocardial infarction | within 180 days
Proportion of participants with vascular death | within 180 days
mRS score collected at 90 days | at 90 days

OTHER OUTCOMES:
Preplanned subgroup analysis | during admission (within 14 days), within 180days
  For the primary endpoint, analyses will be performed in the following subgroups:
  Proportion of occurrence of composite endpoint* in patients with
  1. Intracranial atherosclerosis
  2. Extracranial atherosclerosis
  3. Stent insertion
  4. CYP2C19 poor metabolizers
     * Composite endpoint: Neurologic deterioration during admission (within 14 days) or recurrence of ischemic stroke within 180 days after stroke
Time to recurrence of ischemic stroke | within 180days

CONTACTS AND LOCATIONS:
Locations (24):
- South Korea (24):
  - Asan Medical Center, Seoul, Songpa-gu
  - Pusan National University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Chilgok Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Eulji University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Hallym University Medical Center, Gyeonggi-do
  - Hanyang University Guri Hospital, Gyeonggi-do
  - Korea University Ansan Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Jeju National University Hospital, Jeju City
  - Jeonbuk National University Hospital, Jeonju
  - Ewha Womans University Seoul Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Kyung Hee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Yonsei University Health System, Gangnam Severance Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No